CLINICAL TRIAL: NCT01711905
Title: Study on the Effects of a Recommendation Based Supply of Vitamin D3 in Healthy Volunteers - a Randomized Trail
Brief Title: Study on the Effects of a Recommendation Based Supply of Vitamin D3 in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Ulrike Lehmann, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0315668
Record Dates: First submitted 2012-10-15; First posted 2012-10-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Deficiency of Vitamin D3
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): cholecalciferol 20 µg per day for 12 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (No Intervention): Placebo for 12 weeks

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — daily dosage of 20 µg Vitamin D3 for 12 weeks
  Other Names: cholecalciferol
  Arms: Vitamin D3

SUMMARY:
The aim of this study is to investigate whether a supplementation of 20 µg Vitamin D3 per day for 12 weeks can be used to normalize vitamin d-Status

DETAILED DESCRIPTION:
It is the objective of this study to investigate whether a supplementation with Vitamin D3 can be used to normalize insufficient vitamin d status and reduce atherosclerotic risk factors such as hypertension, inflammation and hyperlipidemia. The research question is whether Vitamin D3 reduces the level of systemic inflammation and whether Vitamin D3 has an effect on blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age between 18 and 70 years
* informed consent

Exclusion Criteria:

* use of antihypertensive medication
* use of vitamin d or calcium supplements
* known renal, inflammatory or malignant diseases
* hypercalcemia or hypercalciuria
* participation in other clinical studies
* use of tanning booths during the study
* pregnancy or lactating period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D3 | after 12 weeks of supplementation
  major outcome variable is the increase of 25-hydroxyvitamin D3 in the treatment group in comparison with the placebo group

SECONDARY OUTCOMES:
atherosclerotic risk factors | after 12 weeks of supplementation
  It is the objective of this study to investigate whether a supplementation with Vitamin D3 can be used to reduce atherosclerotic risk factors such as hypertension, inflammation and hyperlipidemia. The research question is whether Vitamin D3 can reduces the level of systemic inflammation and whether Vitamin D3 has an effect on blood lipids.
inflammation | after 12 weeks of supplementation
  It is the objective of this study to investigate whether a supplementation with Vitamin D3 can be used to reduce inflammation as an atherosclerotic risk factor
hyperlipidemia | after 12 weeks of supplementation
  It is the objective of this study to investigate whether a supplementation with Vitamin D3 can be used to reduce hyperlipidemia as an atherosclerotic risk factor

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele I Stangl, Prof. Dr., Study Director — Institut für Agrar- und Ernährungswissenschaften
Locations (1):
- Naturwissenschaftliche Fakultät III, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Derived] Lehmann U, Riedel A, Hirche F, Brandsch C, Girndt M, Ulrich C, Seibert E, Henning C, Glomb MA, Dierkes J, Stangl GI. Vitamin D3 supplementation: Response and predictors of vitamin D3 metabolites - A randomized controlled trial. Clin Nutr. 2016 Apr;35(2):351-358. doi: 10.1016/j.clnu.2015.04.021. Epub 2015 May 19. PMID 26037521